CLINICAL TRIAL: NCT03319108
Title: The Effect of Severity of Co-morbidity on Outcomes of Pulmonary Rehabilitation in Chronic Obstructive Pulmonary Disease Patients
Brief Title: Comorbidity and Pulmonary Rehabilitation in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Asst. Prof., Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IzmirKCU5
Record Dates: First submitted 2017-10-19; First posted 2017-10-24 (Actual); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Comorbidity Index Score (Other): CCI; 1-3 as Group 1
  Interventions: Other: Exercise
- High Comorbidity Index Score (Other): CCI; 4 and above as Group 2
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Pulmonary Rehabilitation Program for 8 weeks

SUMMARY:
Our aim in this study is to determine the distribution of comorbidity in patients with COPD participating in the pulmonary rehabilitation program and to examine the effect of severity of comorbidy on pulmonary rehabilitation outcomes.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease (COPD) is associated not only with respiratory system effects but also with systemic outcomes leading to numerous chronic comorbidities, and it is well known that patients benefit from pulmonary rehabilitation programs. However, the effect of presence of comorbidity on the outcome of pulmonary rehabilitation in patients with COPD is not clear. Therefore, our aim in this study is to determine the distribution of comorbidity in patients with COPD participating in the pulmonary rehabilitation program and to examine the effect of severity of comorbidy on pulmonary rehabilitation outcomes We included a total of 173 patients referred to the Izmir Suat Seren Chest Diseases and Surgery Training and Research Hospital Pulmonary Rehabilitation Unit. Comorbidities were recorded based on self reports. Charlson Comorbid Indexes (CCI) were calculated. Patients who defined at least one comorbidity were divided into two groups according to CCI; 1-3 as Group 1 and 4 and above as Group 2. Six minute walk test, mMRC dyspnea scale, SGRQ Respiratory Disease Questionnaire, respiratory function tests and arterial blood gases performed for assessment of patients before and after 16 sessions of pulmonary rehabilitation program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Above 18 years
Enrollment: 173 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | 6 minute
  Six minute walk test

SECONDARY OUTCOMES:
Respiratory Functions | 30 minutes
  Pulmonary Function Tests
Dyspnea | 5 minutes
  MMRC dyspnea scale
Disease Specific Quality of Life | 20 minutes
  St George Respiratory Questionnaire
Health Related Quality of Life | 20 minutes
  SF-36

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Naz I, Sahin H, Varol Y, Komurcuoglu B. The effect of comorbidity severity on pulmonary rehabilitation outcomes in chronic obstructive pulmonary disease patients. Chron Respir Dis. 2019 Jan-Dec;16:1479972318809472. doi: 10.1177/1479972318809472. PMID 30428708